CLINICAL TRIAL: NCT01088191
Title: Phase 2 Study to Assess Safety & Tolerability of a Single Injection Into the Knee Joint of Two Different Doses of MSB-CAR001 Combined With Hyaluronan Compared to Hyaluronan Alone in Patients Who Have Undergone an ACL Reconstruction
Brief Title: Safety and Efficacy Study of MSB-CAR001 in Subjects 6 Weeks Post an Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSB-CAR001
Record Dates: First submitted 2010-03-11; First posted 2010-03-17 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Anterior Cruciate Ligament Injury; Osteoarthritis
Keywords: Acute Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Reconstruction; Adult Stem Cells; Mesenchymal precursor cells
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis | interventions — Hyaluronic Acid; Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyaluronan Alone (Active Comparator): Hyaluronan Alone
  Interventions: Biological: MSB-CAR001 Combined With Hyaluronan; Drug: Hyaluronan
- MSB-CAR001 (Experimental): Single Dose of MSB-CAR001 Combined With Hyaluronan
  Interventions: Biological: MSB-CAR001 Combined With Hyaluronan

INTERVENTIONS:
Biological: MSB-CAR001 Combined With Hyaluronan — Knee Injection of Biological: MSB-CAR001 Combined With Hyaluronan
  Single Injection Into the Knee Joint of Single Doses of MSB-CAR001 Combined With Hyaluronan
  Other Names: Anterior Cruciate Ligament Reconstruction; Adult Stem Cells; Knee Injection
Drug: Hyaluronan — Hyaluronan alone
  Other Names: Active Control
  Arms: Hyaluronan Alone

SUMMARY:
The purpose of this study is to evaluate safety and preliminary efficacy of MSB-CAR001 in subjects who have recently undergone an Anterior Cruciate Ligament Reconstruction

DETAILED DESCRIPTION:
This is a prospective, single center, randomized, double blind, controlled Phase 1b/2a study designed to evaluate the safety and tolerability of a single injection into the knee joint of two different doses of MPCs combined with Hyaluronan compared to Hyaluronan alone in patients who have recently undergone an Anterior Cruciate Ligament Reconstruction.

All subjects in this study have undergone unilateral ACL reconstruction surgery within six months of injury. MSB-CAR001 plus Hyaluronan at one of two doses or Hyaluronan alone will be injected into the knee joint.

After the screening and injection visits, each subject will be evaluated clinically within 3 days and 28 days after surgery, and at 2, 3, 6, 9, 12, 18, and 24 months after surgery. The radiographical exams will be performed at 6, 12, 18, and 24 months after surgery.

Subjects will be evaluated at 24 months after surgery for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18 years of age, but not older than 40
2. ACL injury requiring reconstruction
3. Have undergone unilateral ACL reconstruction surgery within six months of injury;
4. Willing and able to undertake a standardized rehabilitation protocol
5. ACL graft used is autograft
6. Willingness to participate in follow-up for 24 months from the time of initial treatment
7. Ability to understand and willingness to sign consent form

Exclusion Criteria:

1. Women who are pregnant or breast feeding or planning to become pregnant during the study
2. Previous allergic reaction to Hyaluronan
3. Systemic or local infection at the screen visit or at the time of the study injection
4. History of any autoimmune disease, such as, systemic lupus erythematosus, Addison's disease, Crohn's disease, or rheumatoid arthritis
5. Treatment with immunosuppression therapy within 6 months prior to screen (visit 1)
6. Acute or chronic infectious disease, including but not limited to human immunodeficiency virus (HIV);
7. Treatment and /or uncompleted follow-up treatment of any investigational therapy within 6 months before the procedure and /or intent to participate in any other investigational drug or cell therapy study during the 24 month follow-up period of this study;
8. Recipient of prior allogeneic stem cell/progenitor cell therapy
9. Undergoing a simultaneous procedure to the opposite knee
10. 20% or greater anti-human leukocyte antigen (HLA) antibody titer and/or has antibody specificities to donor HLA antigens;
11. Known sensitivities to bovine (cow), murine (mouse), chicken products and/or dimethylsulfoxide (DMSO). Previous allergic reaction to Hyaluronan;
12. History or current evidence of alcohol or drug abuse or is a recreational user of illicit drugs or prescription medications
13. History of prior surgery to the study knee joint
14. History of malignancy (excluding basal cell carcinoma that has been successfully excised)
15. Chondral lesions noted at time of surgical reconstruction greater than Grade 1a on any surfaces

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2013-11 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To determine the overall safety of MSB-CAR001 plus carrier using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests (hematology, serum chemistry, inflammation, and immunology). | 2 years

SECONDARY OUTCOMES:
To evaluate the overall efficacy with MSB-CAR001 plus Hyaluronan compared to Hyaluronan alone using MRI scans and x-ray of the involved knee joint and access the change in outcomes (KOOS, SF-36) and pain (VAS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Donna Skerrett, MD, Study Director — Mesoblast, Ltd.
Locations (1):
- Emeritus Research, Malvern East, Victoria, Australia

REFERENCES:
- [Derived] Wang Y, Shimmin A, Ghosh P, Marks P, Linklater J, Connell D, Hall S, Skerrett D, Itescu S, Cicuttini FM. Safety, tolerability, clinical, and joint structural outcomes of a single intra-articular injection of allogeneic mesenchymal precursor cells in patients following anterior cruciate ligament reconstruction: a controlled double-blind randomised trial. Arthritis Res Ther. 2017 Aug 2;19(1):180. doi: 10.1186/s13075-017-1391-0. PMID 28768528
- See also: Sponsor Website — http://www.mesoblast.com